CLINICAL TRIAL: NCT01335555
Title: The Effect of Neoadjuvant Chemotherapy on Lactate Threshold in Patients With Surgically Resectable Upper Gastrointestinal Cancer.
Brief Title: The Effect of Chemotherapy on Lactate Threshold in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: MS. Michelle Mossa, Aintree University Hospitals NHS Foundation Trust
Other Study IDs: 08/H1001/137
Record Dates: First submitted 2011-04-11; First posted 2011-04-14 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2007-08

CONDITIONS: Effects of Chemotherapy; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Pre and Post-chemotherapy

SUMMARY:
It is important to assess patients' fitness for major cancer surgery which carries a high risk of mortality. Patients with poor heart and lung function have a higher risk of death after major cancer surgery. Cardiopulmonary exercise testing, CPET, is an objective measure of patients' fitness. Most patients, before surgery to resect their cancer, undergo a period of chemotherapy. Chemotherapy often regresses the cancer but also has adverse effects on cell function. Our hypothesis is that chemotherapy alters patient fitness, as assessed by CPET, prior to major cancer surgery. Participating patients will undergo fitness testing by CPET before and after their chemotherapy, prior to their surgery.

DETAILED DESCRIPTION:
Purpose: To evaluate the effects of chemotherapy on pre-operative fitness of patients prior to major cancer surgery.

Design: Patients will act as their own case-control.

Patients will be consented at the earliest available opportunity following the decision that they have surgically treatable disease and they consent to pre-operative NAC. Consent for the study will be gained as an outpatient. At "visit 1" patients will undergo CPET, as is our current standard practice, prior to commencing neoadjuvant chemotherapy. As part of the assessment, they will have pulmonary function testing (static lung volumes, lung diffusing capacity),and a nutritional assessment using bioimpedance measurements. They will then undergo 3 cycles of NAC lasting a total of 6 weeks, as is standard current practice at our institution. At "visit 2", approximately four to six weeks following chemotherapy and just prior to planned surgery the CPET and other assessments will be repeated. This is also current standard practice at our institution.

Data from visit 1 and visit 2 will be compared in a paired manner. A statistician will be consulted to assess the degree of normality of the data, the statistical tests to use, and for power calculations. At no point will any treatments be postponed or changed solely for the purposes of collecting data for the research. 12 months survival will be assessed as an outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients with surgically resectable oesophageal and gastric cancers referred to a tertiary NHS referral service who are deemed by their clinician to be suitable for pre-operative neoadjuvant chemotherapy(NAC)prior to their planned surgery.

Exclusion Criteria:

* Patients with cancers deemed to have surgically non-resectable disease, patients refusing chemotherapy, patients unable to perform cardiopulmonary exercise testing (CPET) due to other coincident illness or conditions (e.g. arthritis), patients refusing surgery, patients withholding consent. Patients unable to give informed consent due to mental incapacity. Prisoners will be excluded. Patients in whom haemoglobin drops by >2g/dl between Visit 1 and visit 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Upper gastrointestinal cancer patients receiving neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
What is the effect of chemotherapy on the fitness of patients prior to cancer surgery? | 2 years
  Fitness will be assessed using "cardiopulmonary exercise testing", which is currently a routine part of our clinical practice in pre-operative assessment of patients prior to surgery.

SECONDARY OUTCOMES:
Does good nutritional status following chemotherapy protect against any effect of chemotherapy? | 2 years
Survival outcome at 1 year | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Raw, Principal Investigator — Aintree University Hospitals NHS Foundation Trust, Liverpool, UK
Locations (1):
- Aintree University Hospitals, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Jack S, West MA, Raw D, Marwood S, Ambler G, Cope TM, Shrotri M, Sturgess RP, Calverley PM, Ottensmeier CH, Grocott MP. The effect of neoadjuvant chemotherapy on physical fitness and survival in patients undergoing oesophagogastric cancer surgery. Eur J Surg Oncol. 2014 Oct;40(10):1313-20. doi: 10.1016/j.ejso.2014.03.010. Epub 2014 Mar 27. PMID 24731268